CLINICAL TRIAL: NCT01617785
Title: Patient-centered Evaluative Assessment of Cardiac Events (PEACE): Prospective Study of Patients With Three-vessel Coronary Heart Disease
Brief Title: PEACE Prospective Study of Patients With Three-vessel Disease
Acronym: PEACE3VD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: fuwai201112
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease; Therapeutics; Outcome Assessment
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- CABG group: Three-vessel disease patients undergoing CABG at index hospitalization
- PCI group: Three-vessel disease patients undergoing PCI at index hospitalization
- OMT group: Three-vessel disease patients undergoing no revascularization at index hospitalization

SUMMARY:
Coronary heart disease (CHD) pose a serious health threaten to population. Optimal revascularization strategy in multiple vessel coronary artery disease patients remains a subject of debate between interventional cardiologists and surgeons. Knowledge about the real-life revascularization pattern and outcomes in China is limited. By consecutively recruiting three vessel coronary heart disease patients in 23 geographically representative highest-rank hospitals, this study will examine revascularization strategy, and various real-life factors, that may affect patients lone-term recovery. Practical guidelines, appropriateness criteria and quality evaluative system for revascularization strategy will be established based on the findings, to improve patients outcomes in future finally.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a major concern in public health globally, as well as in China, and remarkable variations of resources available and health system performance have been noted. Relatively limited information is available about how evidence-based therapies are incorporated appropriately into routine clinical practice. Optimal revascularization strategy in multiple vessel coronary artery disease patients remains a subject of debate between interventional cardiologists and surgeons. Practical and applied knowledge from large unselected population is needed to guide practice and policy for quality improvement and cost reduction.

This study will enroll patients with diagnosis of three-vessel disease, or left main disease with significant lesion (over 50%) consecutively in 23 tertiary hospitals scattered all over China. At study entry, participants will be interviewed during their index hospitalization, to collect information about symptoms, functioning, quality of life, and medical care. Demographic characteristics, medical history, clinical features, diagnostic tests, medications, procedures, and in-hospital outcomes of patients will be abstracted from medical records by well trained professional abstractors. And CAG imaging will be reviewed by national and international expert panels. At 1 month, 6 month, and 12 month after discharge, participants will return to the clinic for follow up visits, a face-to-face interview will be conducted to get information about clinical events, symptoms, functioning, quality of life, and medical care during the recovery period. At 1-Month and 12-Month follow-up visit, blood and urine sample will be collected. Participants' blood samples will be stored for future biologic and genetic studies. This study will examine various real-life factors that may affect multiple vessel coronary heart disease patients recovery after PCI/CABG/medications, including patients' characteristics and treatment measures. Practical guidelines, quality evaluative system, and appropriateness criteria will be established based on the findings, to improve patients outcomes in future finally.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized elective patients with diagnosis of three-vessel disease, or left main disease with significant lesion (over 50%), using selective coronary angiography at index hospitalization

Exclusion Criteria:

* Emergent patients, 1-2 vessel disease, Previous CABG or PCI, Combined with other diseases needed cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elective patients for coronary angiogram.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | one year
  Composite of major adverse cardiac events (MACE) including death, myocardial infarction and/or revascularization.

SECONDARY OUTCOMES:
Coronary death or myocardial infarction (fatal or non-fatal MI) | one year
Coronary revascularization procedure | one year
Presumed ischemic stroke (i.e. not known to be hemorrhagic) | one year
Death from all cardiovascular causes | one year
Re-admission | one year
Status of general health (SF-12) | one year
Quality of life (EQ-5D) | one year
Cost-effectiveness | one year

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, M.D., Principal Investigator — National Center for Cardiovascular Diseases; Harlan M Krumholz, M.D., S.M., Principal Investigator — Yale University
Locations (1):
- National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China